CLINICAL TRIAL: NCT05014997
Title: Triglyceride-Glucose Index Levels in Patients With Klinefelter Syndrome and Its Relationship With the Endothelial Dysfunction and Insulin Resistance: A Cross-sectional Observational Study
Brief Title: TyG Index Levels in Klinefelter Syndrome
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, İbrahim Demirci, Dr., Gulhane Training and Research Hospital
Other Study IDs: GMS_21
Record Dates: First submitted 2021-08-16; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Cardiac Event; Klinefelter Syndrome; Endothelial Dysfunction
Keywords: Klinefelter Syndrome, TyG Index, Cardiometabolic risk
MeSH Terms: conditions — Cardiovascular Diseases; Klinefelter Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: 30 male patients with Klinefelter syndrome who were not previously given testosterone replacement.
  Interventions: Other: no intervention
- Control: 30 healthy control subject without diagnosis of any chronic disease
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — this study was designed as retrospective observational study

SUMMARY:
It is well known that the frequency of cardiometabolic diseases are increased in patients with Klinefelter Syndrome. The triglyceride-glucose index (TyG index) is a simple surrogate marker of insulin resistance and is also associated with various cardiometabolic diseases. The aim of this study to investigate the TyG index levels and its relationship with insulin resistance and endothelial dysfunction in patients with KS.

DETAILED DESCRIPTION:
From the patient database of our Endocrinology department we randomly included a total of 30 patients with KS and 32 healthy controls in the study. All the recorded data in the database were registered under the approval of Local Ethical Committee of Gulhane School of Medicine.

The clinical and laboratory parameters, TyG index, asymmetric dimethylarginine (ADMA), homeostatic model assessment of insulin resistance (HOMA-IR) and high-sensitivity C-reactive protein (hs-CRP) levels were gathered from the database and the triglyceride-glucose index was calculated by the help of pre-measured laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a verified Klifelter Syndrome karyotype (all subjects included were 47, XXY) and who were not previously given testosterone replacement.

Exclusion Criteria:

* age <18 years,
* acute infection, malignancy, any visceral organ dysfunction, nutritional derangements, clinical history of cardiovascular disease, cerebrovascular disease, drug use such as antidiabetic or lipid-lowering medications, or those lacking complete clinical data.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We had a patient database consisting of male patients with Klinefelter syndrome
Study Population: A total of 30 male patients with treatment-naive Klinefelter syndrome and 30 control subjects without any chronic disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2013-02-10 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Cardiometabolic risk | 1 day
  Triglyceride - Glucose Index

CONTACTS AND LOCATIONS:
Overall Officials: Alper Sonmez, Prof., Study Director — Health Sciences University, Gulhane School of Medicine, dep. of Endocrinology and Metabolism, Turkey

IPD SHARING:
Plan to Share IPD: No